CLINICAL TRIAL: NCT00581243
Title: An Ascending Multiple-Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of SLV-313 Sustained-Release (SR) Tablets Administered Orally to Subjects With Schizophrenia and Schizoaffective Disorder
Brief Title: Study Evaluating Safety and Tolerability of Ascending Multiple Dose of SLV-313 in Schizophrenia Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 3170A1-01001
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Safety,Tolerability, Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 2 mg SLV-313 SR (fixed dose)
  Interventions: Drug: SLV-313 SR
- 2 (Experimental): 5 mg SLV-313 SR (fixed dose)
  Interventions: Drug: SLV-313 SR
- 3 (Experimental): 10 mg SLV-313 SR (fixed dose)
  Interventions: Drug: SLV-313 SR
- 4 (Experimental): xx mg SLV-313 SR (titration)
  Interventions: Drug: SLV-313 SR

INTERVENTIONS:
Drug: SLV-313 SR — sustained relase tablets taken once daily for 14 days

SUMMARY:
Randomized, inpatient, ascending multiple dose study given to subjects with schizophrenia and schizoaffective disorder to assess safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Men, aged 18-50 years old
* Women, aged 18-50 years old

Exclusion Criteria:

* Non-lactating women, aged 18-50 years old
* Non-pregnant women, aged 18-50 years old

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2008-05-01 (Actual); Study Completion 2008-05-01 (Actual)

PRIMARY OUTCOMES:
Observe safety and tolerability | 25 days

SECONDARY OUTCOMES:
PK and PD profile | 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer